CLINICAL TRIAL: NCT00314106
Title: Phase II Study Using a Myeloablative Lymphocyte Depleting Regimen of Chemotherapy and Intensive Total Body Irradiation Followed by Infusion of Tumor Reactive Lymphocytes and Reconstitution With CD34+ Stem Cells in Metastatic Melanoma
Brief Title: Chemotherapy, Irradiation, Cell Infusions, and Interleukin-2 to Treat Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060136; 06-C-0136; NCT00335127 (obsolete NCT alias)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-09

CONDITIONS: Metastatic Melanoma
Keywords: Clinical Response; Stage IV Melanoma; Adoptive Cell Therapy; Tumor Infiltrating Lymphocytes; Immunologic Response; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Toll-Like Receptor 1; Cyclophosphamide; Interleukin-2; aldesleukin; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBI 1200 cGy + TIL +HD IL-2, prior IL-2 (Experimental): Patients that received prior interleukin 2 (IL-2) therapy will receive a myeloablative lymphocyte depleting preparative regimen consisting of cyclophosphamide (60 mg/kg/day x 2 days intravenous (IV)), fludarabine (25mg/m^2/day IV X 5 days) and 1200 cGy total body irradiation (TBI). Following the lymphodepleting regimen, patient will receive intravenous adoptive transfer of tumor reactive lymphocytes (minimum 3 X 10 (9) and up to a maximum of 3 X 10(11) lymphocytes) followed by high-dose intravenous (IV) IL-2 (720,000 IU/kg/dose every 8 hours for up to 15 doses).
  Interventions: Biological: Melanoma Reactive TIL; Drug: Cyclophosphamide; Biological: IL-2; Drug: Fludarabine; Radiation: 1200 total body irradiation (TBI)
- TBI 1200 cGy + TIL +HD IL-2, no prior IL-2 (Experimental): Patients that have not received prior interleukin 2 (IL-2) therapy will receive a myeloablative lymphocyte depleting preparative regimen consisting of cyclophosphamide (60 mg/kg/day x 2 days intravenous (IV)), fludarabine (25mg/m^2/day IV X 5 days) and 1200 cGy total body irradiation (TBI). Following the lymphodepleting regimen, patient will receive intravenous adoptive transfer of tumor reactive lymphocytes (minimum 3 X 10 (9) and up to a maximum of 3 X 10(11) lymphocytes) followed by high-dose intravenous (IV) IL-2 (720,000 IU/kg/dose every 8 hours for up to 15 doses)
  Interventions: Biological: Melanoma Reactive TIL; Drug: Cyclophosphamide; Biological: IL-2; Drug: Fludarabine; Radiation: 1200 total body irradiation (TBI)

INTERVENTIONS:
Biological: Melanoma Reactive TIL
  Other Names: (TIL) tumor infiltrating lymphocytes
Drug: Cyclophosphamide — 60 mg/kg/ day x 2 days intravenous
  Other Names: Cytoxan
Biological: IL-2 — 720,000 IU/kg/dose every 8 hours for up to 15 doses
  Other Names: Aldesleukin
Drug: Fludarabine — 25 mg/m^2/day intravenous x 5 days
  Other Names: Fludara
Radiation: 1200 total body irradiation (TBI) — 1200 cGY total body radiation
  Other Names: TBI

SUMMARY:
Background:

* In a study in humans with melanoma, patients given total body irradiation to suppress the immune system in conjunction with chemotherapy showed a significant clinical response.
* In previous studies, about one-half of patients given tumor-fighting cells (cells created from the patient's tumor cells and grown in the laboratory) showed some anti-tumor response.

Objective: To determine whether tumor-fighting cells taken from a melanoma tumor and grown in the lab can more effectively at fight melanoma when the patient's immune system is suppressed and cannot attack them.

Eligibility: Patients 18 years of age or older with metastatic melanoma who have tumor reactive cells available.

Design:

-Patients are assigned to one of two groups - those having received prior therapy with Interleukin-2 (IL-2) and those who have not.

After five days of injections of filgrastim, a medicine to stimulated the growth of white blood cells, patients undergo apheresis or bone marrow harvesting, or both, to collect stem cells for later re-infusion. For apheresis, whole blood is collected through a needle in an arm vein and circulated through a cell-separating machine where the stem cells are extracted. The rest of the blood is returned through the same needle or a needle in the other arm. Bone marrow harvesting is done under general anesthesia. Stem cells are collected through a large needle inserted into the hipbone.-Patients' immune system cells and bone marrow function are eliminated with chemotherapy (7 days) and total body irradiation (3 days) so the patient's immune system cells will not fight the tumor-fighting cells they are given in treatment.

* 1 to 3 days after total body irradiation, patients receive the tumor-fighting cells by intravenous (IV) infusion. After the cells are infused, they receive interleukin-2 (IL-2) infusions every 8 hours for 5 days.
* 2 days after infusion of the tumor-fighting cells, patients receive the stem cells collected earlier by apheresis.
* Patients are evaluated 4 to 6 weeks after cell infusion to look for tumor response to treatment. Patients whose tumor has not grown return to the National Institutes of Health (NIH) every 1 to 3 months for blood tests, scans and x-rays.

DETAILED DESCRIPTION:
Background:

The use of immunosuppression prior to adoptive transfer of lymphocytes from tumor bearing mice was based on a variety of murine models demonstrating improved therapeutic effectiveness of the adoptive transfer of lymphocytes following immunosuppression of the host.

Because the degree of immunosuppression has been highly correlated with the ability to eliminate large tumors in murine models, we have been conducting a clinical trial, 04-C-0288, in which 200cGy of total body irradiation is used in conjunction with the same cyclophosphamide and fludarabine regimen used in our prior adoptive cell therapy trials which have demonstrated significant clinical responses.

We have measured T-regulatory cells in patients participating in 04-C-0288 and have demonstrated that despite the addition of 200cGy total body irradiation (TBI), T-regulatory cells promptly reconstituted in the host. Complete clinical responses have not been significantly improved over other adoptive cell therapy regimens.

Thus, in this trial we would like to more adequately test our hypothesis that more intensive lymphodepletion will increase complete responses and persistence of the transferred cells.

Objective:

To determine whether tumor reactive lymphocytes infused in conjunction with the administration of high-dose IL-2 in patients who have received prior therapy with IL-2 and those who have not may result in complete clinical tumor regression in patients with metastatic melanoma receiving a myeloablative lymphoid depleting preparative regimen.

To evaluate the safety of the treatment in patients receiving the myeloablative conditioning regimen, cell transfer and IL-2.

To determine the survival in patients, of infused cells following the administration of the myeloablative regimen, using analysis of the sequence of the variable region of the T cell receptor or flow cytometry (FACS).

Eligibility:

Patients who are greater than or equal to 18 years of age who have tumor reactive cells available, with metastatic melanoma, and are physically able to tolerate high-dose IL-2.

Design:

Patients will be assigned to one of two cohorts, those having received prior therapy with IL-2 and those who have not.

Patients will receive a myeloablative lymphocyte depleting preparative regimen consisting of cyclophosphamide (60 mg/kg/day x 2 days IV), fludarabine (25mg/m^2/day IV X 5 days) and 1200 cGy total body irradiation (TBI).

Patients will receive intravenous adoptive transfer of tumor reactive lymphocytes (minimum 3 X 10 (9) and up to a maximum of 3 X 10(11) lymphocytes) followed by high-dose intravenous (IV) IL-2 (720,000 IU/kg/dose every 8 hours for up to 15 doses).

On day 1 of patients will receive intravenous administration of cryopreserved autologous CD34+ cells.

A complete evaluation of evaluable lesions will be conducted 4-6 weeks after cell infusion. Patients will be enrolled into two strata, using a phase II optimal design to rule out a modest CR rate of 24%, with 33-54 patients enrolled in each strata.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have tumor reactive cells obtained and evaluated while participating in the Surgery Branch protocol, "Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols" or on another Institutional Review Board (IRB) approved Surgery Branch adoptive cell therapy study, i.e. 99-C-0158 or 03-C-0162.

The first ten patients enrolled must have previously received interleukin-2 (IL-2) and have been either non-responders (progressive disease) or have recurred.

Patients must be greater than or equal to 18 years of age and must have measurable metastatic melanoma.

Patients of both genders must be willing to practice birth control during treatment and for four months after receiving the preparative regimen.

Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1.

Absolute neutrophil count greater than 1000/mm^3 without support of filgrastim.

Platelet count greater than 100,000/mm^3.

Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than three times the upper limit of normal.

Serum creatinine less than or equal to 1.6 mg/dl.

Total bilirubin less than or equal to 2 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dl.

Must be willing to sign a durable power of attorney.

Patients must be able to understand and sign the Informed Consent document.

Patients with resected or stable brain metastases will be eligible.

Left ventricular ejection fraction (LVEF) greater than or equal to 45%.

Carbon monoxide diffusing capacity (DLCO) greater than or equal to 60% predicted.

CELL INFUSION EXCLUSION CRITERIA:

Less than 30 days has elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, or less than six weeks since prior nitrosurea therapy. All patients' toxicities must have recovered to a grade 1 or less or as specified in the eligibility criteria. Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria.

Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.

Life expectancy of less than three months.

Systemic steroid therapy required.

Hemoglobin less than 8 g/dl unable to be corrected with transfusion.

Any active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.

Any form of primary or secondary immunodeficiency. Must have recovered immune competence after chemotherapy or radiation therapy as evidenced by normal ANC greater than 1000/mm^3 and absence of opportunistic infections. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)

Seropositive for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)

Patients with hepatitis B or hepatitis C will be excluded.

Seronegative for Epstein-Barr virus (EBV).

Patients who are not willing to complete a durable power of attorney (DPA) will be excluded.

Patients who have received prior preparative regimens with cyclophosphamide and fludarabine on prior Surgery Branch adoptive cell therapies will be excluded.

The following patients will be excluded because of inability to receive high dose IL-2:

Patients will be excluded if they have a history of electrocardiogram (EKG) abnormalities, symptoms of cardiac ischemia or arrhythmias and have a LVEF less than 45% on a cardiac stress test (stress thallium, stress multi-gated acquisition scan (MUGA), dobutamine, echocardiogram or other stress test).

Similarly, patients who are 50 years old or greater with an LVEF less than 45% will be excluded.

Patients who have a prolonged history of cigarette smoking or symptoms of respiratory dysfunction will be excluded if they have an abnormal pulmonary function test as evidenced by a forced expiratory volume 1 (FEV1) less than 60% predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-04; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rooney CM, Smith CA, Ng CY, Loftin S, Li C, Krance RA, Brenner MK, Heslop HE. Use of gene-modified virus-specific T lymphocytes to control Epstein-Barr-virus-related lymphoproliferation. Lancet. 1995 Jan 7;345(8941):9-13. doi: 10.1016/s0140-6736(95)91150-2. PMID 7799740
- [Derived] Yao X, Ahmadzadeh M, Lu YC, Liewehr DJ, Dudley ME, Liu F, Schrump DS, Steinberg SM, Rosenberg SA, Robbins PF. Levels of peripheral CD4(+)FoxP3(+) regulatory T cells are negatively associated with clinical response to adoptive immunotherapy of human cancer. Blood. 2012 Jun 14;119(24):5688-96. doi: 10.1182/blood-2011-10-386482. Epub 2012 May 3. PMID 22555974
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2006-C-0136.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TBI 1200 cGy + TIL +HD IL-2, Prior IL-2 | TBI 1200 cGy + TIL +HD IL-2, no Prior IL-2
Started | 18 | 8
Completed | 18 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TBI 1200 cGy + TIL +HD IL-2, Prior IL-2 | TBI 1200 cGy + TIL +HD IL-2, no Prior IL-2 | Total
Number analyzed (Participants) | 18 | 8 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 8 | 26
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.4 (11.4) | 48.5 (10.6) | 44.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 13 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 7 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 8 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Determine if the combination of high dose aldesleukin, reinfused cells after lymphocyte depleting chemotherapy and 1200 cGy total body irradiation (TBI) is able to be associated with a modest fraction of patients with metastatic melanoma who can experience a complete response to therapy.
  Complete response (CR) is a disappearance of all target lesions.
Time Frame: 33 months
Measure: Number; unit: Participants
Arm/Group | TBI 1200 cGy + TIL +HD IL-2, Prior IL-2 | TBI 1200 cGy + TIL +HD IL-2, no Prior IL-2
Number analyzed (Participants) | 18 | 8
Participants | 7 | 3

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 33 months
Measure: Number; unit: Participants
Arm/Group | TBI 1200 cGy + TIL +HD IL-2, Prior IL-2 | TBI 1200 cGy + TIL +HD IL-2, no Prior IL-2
Number analyzed (Participants) | 18 | 8
Participants | 18 | 8

ADVERSE EVENTS:
Arm/Group | TBI 1200 cGy + TIL +HD IL-2, Prior IL-2 | TBI 1200 cGy + TIL +HD IL-2, no Prior IL-2
Serious Adverse Events (participants affected / at risk) | 7/18 | 4/8
Other Adverse Events (participants affected / at risk) | 18/18 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI 1200 cGy + TIL +HD IL-2, Prior IL-2 (N=18) | TBI 1200 cGy + TIL +HD IL-2, no Prior IL-2 (N=8)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 2 (2)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
peripheral nerve infection (Infections and infestations) | 2 (2) | 0 (0)
Bilirubin increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gait abnormal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (General disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI 1200 cGy + TIL +HD IL-2, Prior IL-2 (N=18) | TBI 1200 cGy + TIL +HD IL-2, no Prior IL-2 (N=8)
Autoimmune disorder (Immune system disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 (13) | 5 (7)
Leukocyte count decreased (Blood and lymphatic system disorders) | 17 (20) | 8 (10)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 18 (27) | 8 (12)
Neutrophil count decreased (Blood and lymphatic system disorders) | 17 (18) | 8 (11)
Platelet count decreased (Blood and lymphatic system disorders) | 16 (17) | 8 (8)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 10 (13) | 1 (1)
Fever (General disorders) | 4 (4) | 0 (0)
Insomnia (General disorders) | 2 (2) | 0 (0)
Weight loss (Gastrointestinal disorders) | 5 (5) | 6 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (11) | 4 (4)
Nausea (Gastrointestinal disorders) | 12 (13) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (8) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 10 (10) | 6 (6)
Catheter-related infection (Infections and infestations) | 2 (2) | 0 (0)
vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Edema limbs (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 9 (10) | 5 (5)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Bilirubin increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
serum calcium decreased (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Creatinine increased (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 6 (10) | 4 (5)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Confusion (Nervous system disorders) | 5 (5) | 5 (5)
Euphoria (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain (General disorders) | 3 (4) | 1 (1)
Bone pain (General disorders) | 2 (2) | 0 (0)
Pain in extremity (General disorders) | 3 (4) | 0 (0)
joint pain (General disorders) | 1 (1) | 0 (0)
scrotal pain (General disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 4 (4) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Petechiae (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No